CLINICAL TRIAL: NCT04222439
Title: Development and Validation of a Deep Learning Algorithm for the Diagnosis of Gastrointestinal Diseases
Brief Title: Deep Learning Algorithm for the Diagnosis of Gastrointestinal Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-SDU-QILU-G710
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Gastrointestinal Disease
Keywords: Deep Learning; Central Neural Networks; Endoscopy; Gastrointestinal Disease
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI monitoring gastrointestinal endoscopy (Experimental): After receiving standard preparation regimen, patients go through colonoscopy or gastroscopy under the AI monitoring device. The whole procedure is monitored by AI associated recognition system. Gastrointestinal diseases will be detect and diagnosis in which the AI device will automatically captured relevant images and report the site of each segment on the screen. Histology analysis is set as a golden standard. Then all the AI captured images will be reviewed by human group, which consists of three to five experienced endoscopic physicians.
  Interventions: Device: AI for the Diagnosis of Gastrointestinal Diseases

INTERVENTIONS:
Device: AI for the Diagnosis of Gastrointestinal Diseases — After receiving standard preparation regimen, patients go through colonoscopy or gastroscopy under the AI monitoring device. The whole procedure is monitored by AI associated recognition system. Gastrointestinal diseases will be detect and diagnosis in which the AI device will automatically captured relevant images and report the site of each segment on the screen. Histology analysis is set as a golden standard. Then all the AI captured images will be reviewed by human group, which consists of three to five experienced endoscopic physicians.

SUMMARY:
The purpose of this study is to develop and validate a deep learning algorithm for the diagnosis of gastrointestinal diseases. Then, evaluate the accuracy this new artificial intelligence(AI) assisted recognition system in clinic practice.

DETAILED DESCRIPTION:
Recently, deep learning algorithm based on central neural networks (CNN) has shown multiple potential in computer-aided detection and computer-aided diagnose of gastrointestinal lesions. However, there is still a blank in recognition of all gastrointestinal diseases. This study aim to develop and validate a deep learning algorithm for the diagnosis of gastrointestinal diseases. Then, evaluate the accuracy this new artificial intelligence(AI) assisted recognition system in clinic practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants, aged 18 years or older, who had not had a previous endoscopy were retrieved from all participating hospitals.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
The diagnostic accuracy of gastrointestinal diseases with deep learning algorithm. | 1 month
  The diagnostic accuracy of gastrointestinal diseases with deep learning algorithm.

SECONDARY OUTCOMES:
The diagnostic sensitivity of gastrointestinal diseases with deep learning algorithm. | 1 month
  The diagnostic sensitivity of gastrointestinal diseases with deep learning algorithm.
The diagnostic specificity of gastrointestinal diseases with deep learning algorithm. | 1 month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm.
The diagnostic positive predictive value of gastrointestinal diseases with deep learning algorithm. | 1 month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm.
The diagnostic negative predictive value of gastrointestinal diseases with deep learning algorithm. | 1month
  The diagnostic specificity of gastrointestinal diseases with deep learning algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China